CLINICAL TRIAL: NCT01035125
Title: A Study of Effect of One Week Self-management Program in Patients With Fibromyalgia
Brief Title: Effect of One Week Self-management Program in Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Revmatismesykehuset AS (Other)
Responsible Party: Study chair: Knut Mikkelsen, Revmatismesykehuset AS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: REK 39-07138b 1.2007.1416
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-07

CONDITIONS: Fibromyalgia
Keywords: Self-management; Self-efficacy; Coping; Health consumer; Patient education; Health related quality of life
MeSH Terms: conditions — Fibromyalgia | interventions — Self-Management; Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Waiting list (No Intervention)
- Self-management program (Experimental): One week self-management program
  Interventions: Behavioral: Self-management program

INTERVENTIONS:
Behavioral: Self-management program — Participants will receive a one week inpatient self-management program
  Other Names: Patient education
  Arms: Self-management program

SUMMARY:
The purpose of this study is to explore the effect of one week inpatient self-management program (SMP) in patients with fibromyalgia. The SMP is delivered as group education/activities by allied health professionals.

DETAILED DESCRIPTION:
This study will determine if one week inpatient SMP can reduce FM symptoms and increase patients self-efficacy, health status, quality of life and being active health consumers.

The one-week SMP is designed to help people manage their rheumatic disease and challenges in daily life. The program has the same core concepts as outpatient programmes and comprises information, discussions on how to cope with the disease and daily life, cognitive management skills, exercise, engagement in self-care and interactions with healthcare professionals. During the program, the inpatient education unit takes up to 16 patients and 5 relatives per week within one diagnostic group. Each educational session lasts for 1.5-2.5 hours and the physical activity sessions for 0.5-1 hour. In the evening group sessions, the patients are divided into small groups of approximately five participants. They talk together for one hour under leadership of one health professional who is educated in coaching. The focus is on coping with the disease and daily life.

For the intervention group there will be a one year follow up study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Fibromyalgia outlined by the American College of Rheumatology for one year or more
* Between 20 and 70 years old
* Native Norwegian speaking
* Own wishes about participating the self-management program

Exclusion Criteria:

* Participated in the hospitals' SMP before
* Cognitive dysfunction
* Problems with sight and hearing that not can be compensated
* Mental disorders except light or treated depressions

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2008-12; Primary Completion 2011-02 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
EC-17 (Effective Musculoskeletal Consumer Scale) | Baseline, 3 weeks before the program, 3 weeks and 6 months after the program
GHQ20 (General Health Questionnaire) | Baseline, 3 weeks before the program, 3 weeks and 6 months after the program

SECONDARY OUTCOMES:
FIQ (Fibromyalgia Impact Questionnaire) | Baseline, 3 weeks before the program, 3 weeks and 6 months after the program
SF-36 (Short Form Health Survey) | Baseline, 3 weeks before the program, 3 weeks and 6 months after the program
Self-efficacy Scale | Baseline, 3 weeks before the program, 3 weeks and 6 months after the program

CONTACTS AND LOCATIONS:
Overall Officials: Knut Mikkelsen, MD, Study Chair — Revmatismesykehuset AS, Lillehammer, Norway
Locations (1):
- Lillehammer Hospital for Rheumatic Diseases, Lillehammer, Oppland, Norway

REFERENCES:
- [Derived] Hamnes B, Mowinckel P, Kjeken I, Hagen KB. Effects of a one week multidisciplinary inpatient self-management programme for patients with fibromyalgia: a randomised controlled trial. BMC Musculoskelet Disord. 2012 Sep 26;13:189. doi: 10.1186/1471-2474-13-189. PMID 23013162